CLINICAL TRIAL: NCT04090619
Title: Frequency of Cachexia in Ambulatory Cancer Patients and Psychological Burden in Both Patients and Their Primary Caregivers Who Are Referred to an Outpatient Supportive Care Clinic
Brief Title: Frequency of Cachexia in Ambulatory Cancer Patients and Psychological Burden in Patients and Their Primary Caregivers
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2019-0203; NCI-2019-04590 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0203 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-08-05; First posted 2019-09-16 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Advanced Malignant Solid Neoplasm; Caregiver; Metastatic Malignant Solid Neoplasm; Recurrent Leukemia; Recurrent Lymphoma; Recurrent Malignant Solid Neoplasm; Recurrent Plasma Cell Myeloma
MeSH Terms: conditions — Neoplasm Metastasis; Leukemia; Lymphoma; Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (questionnaires): Participants complete 8 questionnaires about appetite, quality of life, symptoms, history of weight loss, nutritional status, body image, and nutritional support over 30 minutes.
  Interventions: Other: Questionnaire Administration

INTERVENTIONS:
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This trial studies the frequency of cachexia in ambulatory cancer patients and the psychological burden in patients and their primary caregivers who are referred to an outpatient supportive care clinic. Studying how often loss of appetite and/or unintentional weight loss (cachexia) occurs in patients seen in the supportive care clinic may help researchers develop new ways to lower stress in patients who suffer from loss of appetite and weight loss as well as their family caregivers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the proportion of patients with cancer cachexia, as defined by various criteria including The European Society of Clinical Nutrition and Metabolism (ESPEN) as well as an International Consensus Criteria (ICC), in a group of ambulatory patients with advanced cancer who are referred to a Supportive Care Clinic at University of Texas MD Anderson Cancer Center (UTMDACC).

SECONDARY OBJECTIVES:

I. To estimate the proportion of patients with complications anorexia (Appetite Score Edmonton Symptom Assessment Scale [ESAS] [>= 3] & Functional Assessment of Anorexia Therapy-Anorexia/Cachexia Subscale Questionnaire [FAACT-A/CS] =< 37); and the proportion of patients that have both anorexia and cancer cachexia.

II. To examine the association between symptoms of anorexia and/or cancer cachexia and the degree of symptom distress in cancer patients seen in a supportive care clinic, as measured by Edmonton Symptom Assessment Scale (ESAS - total score), Hospital Anxiety and Depression Scale (HADS), and the Functional Assessment of Anorexia Therapy-Anorexia/Cachexia Subscale (FAACT-A/CS Questionnaire) and in their primary caregivers, ESAS-Caregiver, Caregiver Quality of Life-Cancer (CQOLC), and Brief Illness Perception (Brief-IPQ) questionnaire.

III. To elucidate the frequency of Nutritional Impact Symptoms (NIS), evaluated by a Patient-Generated Subjective Global Assessment (PG-SGA-SF), and alterations in body composition (Inbody 770 Bio-Impedance Machine) experienced by patients with advanced cancer.

IV. To evaluate the patient's perception of body image, Body Image Scale (BIS), as related to their change in weight and physical appearance due to cachexia in patients with advanced cancer.

V. To evaluate the perception of need for nutritional support in cancer patients seen in a supportive care clinic.

OUTLINE:

Participants complete 8 questionnaires about appetite, quality of life, symptoms, history of weight loss, nutritional status, body image, and nutritional support over 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. [Patient] Patients visiting the Supportive Care Clinic (SCC) for a consultation or a follow up.
2. [Patient] Patients who can identify a primary caregiver.
3. [Patient] Diagnosis of advanced cancer defined as locally advanced, recurrent, or metastatic.
4. [Patient] Be able to read and speak English.
5. [Patient] 18 years of age or older.
6. [Caregiver] Be identified or self-identified as a primary caregiver of the patient.
7. [Caregiver] Provide informed consent
8. [Caregiver] Be able to read and speak English.
9. [Caregiver] 18 years of age or older.
10. [Caregiver] Caregivers who are not able to complete the questionnaire on the day of patients' SCC visit must be willing to engage in a telephone questionnaire with research staff within 60 days of the patient's enrollment.

Exclusion Criteria:

1. [Patient] Refusal to participate in this study. This study requires both patient and caregiver enrollment.
2. [Patient] Patients with no caregiver or only paid caregivers.
3. [Patient] Patients with cognitive impairment as identified by research staff, treating physician or nurse (Memorial Delirium Assessment Scale score of >/= 7).
4. [Caregiver] Refusal to participate in this study. This study requires both patient and caregiver enrollment.
5. [Caregiver] Not a primary caregiver or is a paid caregiver.
6. [Caregiver] Evidence of cognitive impairment, as determined based on orientation questions pertaining to the date, day of the week, time, and place

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with advanced cancer or relapsed hematological malignancies and their primary caregiver
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Cancer Cachexia | Day 1
  Assessed by either European Society for Clinical Nutrition and Metabolism (ESPEN) includes body mass index (BMI) < 18.5 (mandatory) or combined finding of unintentional weight loss (mandatory) and at least one of either reduced BMI or a low fat free mass index (FFMI), or International Consensus Criteria (ICC) defined as cachexia weight loss greater than 5% over 6 month period or weight loss greater than 2% showing depletion according to current bodyweight and height over an indefinite time point.

SECONDARY OUTCOMES:
Functional Assessment of Anorexia Therapy-Anorexia/Cachexia Subscale Questionnaire (FAACT-A/CS) | Day 1
  For assessment of decreased appetite. Total score ranges from 0 to 48, lower scores indicate decrease appetite.
Hospital Anxiety and Depression Scale (HADS) for assessment of depression and anxiety | Day 1
  A validated tool consists of 14 items scored from 0 to 3 for a total score of 0 to 21. A cut-off score of 8 out of 21 will be used.
Edmonton Symptom Assessment Scale (ESAS) | Day 1
  Edmonton Symptom Assessment Scale ESAS is a validated tool for regular assessment of symptom distress. Grading severity of patient symptoms from "no" 0 to "worst symptom" 10 in the last 24 hours.
Caregiver Quality of Life-Cancer (CQOLC) Questionnaire | Day 1
  Caregiver Quality of Life-Cancer CQOLC is a 35 item cancer-specific instrument that assesses the quality of life of caregiver. Score range from 0-140, with higher scores to reflect better wellbeing.
Brief Illness Perception Questionnaire (IPQ) score | Day 1
  Illness Perception Questionnaire IPQ is a validated self-report to assess perceptions of patient's illness. Each item is scored from 0-10, A higher score reflects a threatening view of illness.
Patient-Generated Subjective Global Assessment (PG-SGA-SF) | Day 1
  Patient-Generated Subjective Global Assessment PG-SGA-SF is a tool used to measure risks for malnutrition. The total score of 4 boxes are calculated, a higher score places patients at a higher risk for developing weight loss.
Body Image Scale (BIS) | Day 1
  Body Image Scale BIS is a validated 10-item scale used to assess body image changes in cancer patients. Each item is answered either "not at all", "a little", "quite a bit", or "very much", scoring as 0 to 3. Higher scores indicate body image dissatisfaction.
Perception of need for nutritional support | Day 1
  is a survey of 3 questions to describe patients' opinions about nutritional support. And evaluates the perception of need for intervention regarding nutrition and interventions for weight loss.

CONTACTS AND LOCATIONS:
Overall Officials: Rony Dev, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org